CLINICAL TRIAL: NCT05376618
Title: Pilot Study on Proteomics of Erythrocyte Proteins in Patients With Chronic Obstructive Pulmonary Disease Based on TMT Technology
Brief Title: Pilot Study on Proteomics of Erythrocyte Proteins in Patients With COPD Based on TMT Technology
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-KY-060--01
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2021-07

CONDITIONS: Protein; Disease
Keywords: copd; erythrocyte; proteomics
MeSH Terms: conditions — Disease; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stable COPD
  Interventions: Other: no intervention
- Healthy
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Chronic obstructive pulmonary disease (COPD), a common and complex disease characterized by persistent airflow limitation, is a leading cause of mortality worldwide. COPD and its comorbidity are associated with hypoxia condition. Further investigations on the cellular and molecular aspects of hypoxia in COPD should help to reveal the mechanisms underlying the development of this disease. Dysfunction of the erythrocyte, a main medium to transport oxygen through the blood, contributes to the prognosis and severity of COPD through hypoxia. It is proposed that dysregulated proteins in erythrocytes that impair oxygen transport may be involved in the development of COPD. However, a comprehensive study on altered proteins of erythrocytes in COPD is still lacking. Proteomics techniques and protein chip techniques provide a high throughput screening method to figure out characteristic inflammatory or metabolic markers of diseases. Therefore, this study is to evaluate the clinical significance of differential erythrocyte proteins in the course of COPD disease.

ELIGIBILITY:
1. case group

   Inclusion Criteria:
   1. Age from 40 to 80 years old; gender is not limited.
   2. Stable COPD
   3. Sign the informed consent with the willingness of obeying the protocol. -

   Exclusion Criteria:
   1. Subjects with known other chronic respiratory diseases except for COPD (such as asthma, tuberculosis, bronchiectasis, interstitial lung disease, occupational lung diseases, sarcoidosis, lung cancer, et al);
   2. Subjects had been accepted lung lobectomy or transplantation;
   3. Subjects be ill with severe, or uncontrolled systemic diseases other than COPD (such as psychiatry diseases, chronic liver diseases, heart failure, auto-immunity diseases, chronic renal diseases, et al );
   4. Alcoholism, drug or solvents addition;
   5. Acute exacerbation COPD patients (AECOPD) -
2. control group Inclusion criteria

   1. Age from 40 to 80 years old; gender is not limited.
   2. Sign the informed consent with the willingness of obeying the protocol. - Exclusion criteria

   <!-- -->

   1. Subjects with known other chronic respiratory diseases (such as COPD, asthma, tuberculosis, bronchiectasis, interstitial lung disease, occupational lung diseases, sarcoidosis, lung cancer, et al);
   2. Subjects had been accepted lung lobectomy or transplantation;
   3. Subjects be ill with severe, or uncontrolled systemic diseases other than COPD (such as psychiatry diseases, chronic liver diseases, heart failure, auto-immunity diseases, chronic renal diseases, et al );
   4. Alcoholism, drug or solvents addition;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be an outpatient-based case-control study. 15 stable COPD patients and 15 healthy individuals will be recruited.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Protein biomarkers in erythrocyte predicting rapid decline of lung function | 2021-7-15 to 2022-7-15
  The study is to identify the biomarkers and make sure which is associated with rapid decline of lung function. The study will include a total of 30 study subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided